CLINICAL TRIAL: NCT00591630
Title: Zevalin/BEAM/Rituximab vs BEAM/Rituximab With or Without Rituximab Maintenance in Autologous Stem Cell Transplantation for Diffuse Large B-Cell Lymphomas
Brief Title: Zevalin/BEAM/Rituximab vs BEAM/Rituximab With or Without Rituximab in Autologous Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-1018; NCI-2012-01753 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Diffuse Large Cell Lymphoma; Lymphoma
Keywords: Diffuse Large Cell Lymphoma; Lymphoma; Zevalin; Ibritumomab; IDEC-Y2B8; Carmustine; BCNU; BiCNU; Etoposide; VePesid; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride; Melphalan; Rituximab; Rituxan; BEAM
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — ibritumomab tiuxetan; Carmustine; Etoposide; Cytarabine; Melphalan; Rituximab; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Zevalin + BEAM + Rituximab +Stem Cell Transplant + Rituximab (Active Comparator): Zevalin + BEAM + Rituximab Followed by Stem Cell Transplant and Maintenance Rituximab
  Interventions: Drug: Zevalin; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Drug: Rituximab; Procedure: Stem Cell Transplant
- Zevalin + BEAM + Rituximab +Stem Cell Transplant (Active Comparator): Zevalin + BEAM + Rituximab Followed by Stem Cell Transplant
  Interventions: Drug: Zevalin; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Drug: Rituximab; Procedure: Stem Cell Transplant
- BEAM + Rituximab + Stem Cell Transplant + Rituximab (Active Comparator): BEAM + Rituximab Followed by Stem Cell Transplant and Maintenance Rituximab
  Interventions: Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Drug: Rituximab; Procedure: Stem Cell Transplant
- BEAM + Rituximab + Stem Cell Transplant (Active Comparator): BEAM + Rituximab Followed by Stem Cell Transplant
  Interventions: Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Drug: Rituximab; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Zevalin — (111In Zevalin) 5 millicurie (mCi) by vein and (90Y Zevalin) 0.4 mCI/kg by vein.
  Other Names: Ibritumomab; IDEC-Y2B8
  Arms: Zevalin + BEAM + Rituximab +Stem Cell Transplant; Zevalin + BEAM + Rituximab +Stem Cell Transplant + Rituximab
Drug: Carmustine — 300 mg/m^2 by vein.
  Other Names: BCNU; BiCNU
Drug: Etoposide — 200 mg/m^2 by vein every 12 hours.
  Other Names: VePesid
Drug: Cytarabine — 200 mg/m^2 by vein every 12 hours.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrocholoride
Drug: Melphalan — 140 mg/m^2 by vein.
Drug: Rituximab — Arm 1, Arm 2 = 250 mg/m^2 by vein;
  Arm 1, Arm 2, Arm 3, Arm 4 = 1000 mg/m^2 by vein following Stem Cell Transplant;
  Arm 1, Arm 3 = 375 mg/m² by vein Maintenance Therapy.
  Other Names: Rituxan
Procedure: Stem Cell Transplant — Injection of stem cells (Autologous SCT)
  Other Names: Stem Cell Transplantation; SCT

SUMMARY:
The goal of this clinical research study is to learn if the addition of 90Y Zevalin to BEAM chemotherapy (carmustine, etoposide, cytarabine, and melphalan) and rituximab is more effective than the combination of BEAM and rituximab alone in patients with lymphoma who receive a stem cell transplant.

DETAILED DESCRIPTION:
The Study Drugs:

90Y Zevalin is designed to attach to lymphoma cells, and destroy the cells using a radiation particle that is attached to it.

111In Zevalin is like 90Y Zevalin, but the radioactive particle that is attached to it does not kill lymphoma cells. The radioactive particle makes the drug able to be seen inside your body. It is being used in this study to predict how fast the study drug will travel in the body and how long the drug stays in the body.

Carmustine, etoposide, cytarabine, and melphalan (BEAM) are designed to kill lymphoma cells by damaging the cells DNA.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

Study Groups 1 and 2:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. You will have an equal chance of being assigned to each group. Group 1 will receive 90Y Zevalin along with rituximab and BEAM therapy. Group 2 will receive rituximab and BEAM therapy. You and the study staff will know which group you are in.

Study Drug Administration:

If you are in Group 1, you will receive rituximab through a needle in your vein (over 4-5 hours) followed by 111In Zevalin by vein (over 15 minutes). A nuclear scan will be done within the following 40 to 48 hours to see how the drug is traveling through your body.

If intolerable side effects are not shown by the scans, you will receive rituximab (over 4-5 hours) and 90Y Zevalin (over 15 minutes) through a needle in your vein 7 days after the 111In Zevalin infusion.

You will begin BEAM chemotherapy 7 days after the second 90Y Zevalin infusion.

BEAM Chemotherapy:

Both groups will have 7 days of BEAM combination chemotherapy.

* On Day 1, you will receive carmustine through a needle in your vein over 1 hour.
* On Days 2-5 you will receive cytarabine by vein (over 1 hour) followed by etoposide (over 3 hours). Both infusions will be repeated every 12 hours on Days 2-5.
* On Day 6 you will be given melphalan by vein over 30 minutes.
* On Day 7 the stem cells that were collected earlier from you will be given back ("transplanted") through a catheter over 30-45 minutes.
* You will also receive rituximab by vein (over 5-7 hours) on Day 8.

You will receive rituximab (over 4-5 hours) 7 days after the stem cell transplant. You will receive G-CSF by injection once a day starting 7 days after the stem cell transplant until your blood counts return to a normal level. You should stay in the Houston area for about 2-4 weeks after the transplant.

Study Procedures:

At about 1 month after the transplant you will have x-rays, CT scans, and positron emission tomography (PET) scans. You will also have a bone marrow aspirate and biopsy to check the status of the disease.

Blood (about 1 tablespoon) will be drawn once a day while you are in the hospital to check your blood counts.

Blood tests (about 1-2 tablespoons), urine tests, bone marrow collections, and x-rays may be done as needed to track the effects of the transplant.

You will have transfusions of blood and platelets as needed.

Study Groups A and B:

About 1 month after the transplant, you will be randomly assigned (as in the toss of a coin) to 1 of 2 new groups (Group A and Group B). Group A will receive rituximab by vein over 5-7 hours, once every 3 months, starting 3 months after the stem cell transplant. You will receive rituximab for the first 18 months after the stem cell transplant. Group B will not receive rituximab. You will have an equal chance of being in each group.

Follow-up Visits:

You will return to the clinic every 6 months for 5 years to check the status of the disease. The following tests and procedures will be performed:

* Blood (about 1-2 tablespoons) and urine will be collected for routine tests.
* You will have a bone marrow biopsy to check the status of the disease.
* You will have a chest x-ray and a CT scan.
* You will have a PET scan.

Length of Study:

You may stay on study as long as you are benefitting. You will be taken off-study if the disease gets worse or intolerable side effects occur.

This is an investigational study. 90Y-Zevalin is approved by the FDA for relapsed and refractory lymphoma. Its use in this study is investigational. 111In Zevalin, Carmustine, etoposide, cytarabine, melphalan, and Rituximab are all FDA approved and commercially available. However, their use together in this study is also investigational. Up to 50 patients will be take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed CD20-positive B-cell diffuse large cell lymphoma (demonstrated in lymph nodes or bone marrow), chemosensitive (at least PR).
2. Age: up to 18-70 years of age.
3. Prestudy performance status of 0, 1, or 2 according to the WHO.
4. No anti-cancer therapy started within three weeks, prior to study initiation, and fully recovered from all toxicities associated with prior surgery, radiation treatments, chemotherapy, or immunotherapy. No prior rituximab within three weeks of starting therapy.
5. If patients had prior radiation, this should have not involved more than 25% of the bone marrow.
6. Acceptable hematologic status within two weeks prior to patient registration, including: Absolute neutrophil count ({segmented neutrophils + bands} x total WBC) > 1,500/mm³ and platelet counts > 80,000/mm³
7. IRB -approved signed informed consent.
8. Patients determined to have <10% bone marrow involvement with lymphoma within 60 days before study entry as defined by bone marrow aspirates and biopsies.
9. Female patients included must not be pregnant or lactating.
10. Patients should have at least 4-6 x 10^6 CD34+/kg peripheral stem cells collected. Around 1-2 million cells will beheld as back up.
11. Voluntary signed, written IRB-approved informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
12. Men and women of reproductive potential must agree to follow accepted birth control methods for the duration of the study. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

1. Failed stem cell collection of >/= 4x10^6CD34+/kg.
2. Prior radioimmunotherapy.
3. Presence of active CNS lymphoma.
4. Patients with abnormal liver function: total bilirubin > 1.5 mg/dl.
5. Patients with abnormal renal function: serum creatinine > 1.6 mg/dl.
6. Serious nonmalignant disease or infection which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives.
7. Corrected DLCO < 50% and FEV subscript 1 or FVC < 50% predicted.
8. Cardiac EF < 50% by 2-D Echogram.
9. Prior radiation to lungs.
10. Abnormal cytogenetics predictive of secondary cancers, such as -5,-7.
11. Pregnant (Positive Beta HCG test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization) or currently breast-feeding. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
12. Patients with other malignancies diagnosed within 2 years prior to Study entry (except skin squamous or basal cell carcinoma).
13. Active uncontrolled bacterial, viral fungal infections.
14. Major surgical procedure or significant traumatic injury within 4 weeks prior to Study entry.
15. Serious, non-healing wound, ulcer, or bone fracture.
16. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 3 months prior to Study entry.
17. History of Stroke within 6 months.
18. Myocardial infarction within the past 6 months prior to Study Day 1, or has New York Heart Association (NYHA) Class III or IV heart failure or arrythmias, unstable angina, uncontrolled congestive heart failure or arrythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by investigator as not medically relevant.
19. Uncontrolled chronic diarrhea.
20. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-11-14 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 - Zevalin + BEAM + Rituximab +Stem Cell Transplant: Zevalin + BEAM + Rituximab Followed by Stem Cell Transplant and Maintenance Rituximab
  Zevalin: (111In Zevalin) 5 millicurie (mCi) by vein and (90Y Zevalin) 0.4 mCI/kg by vein.
  Carmustine: 300 mg/m^2 by vein.
  Etoposide: 200 mg/m^2 by vein every 12 hours.
  Cytarabine: 200 mg/m^2 by vein every 12 hours.
  Melphalan: 140 mg/m^2 by vein.
  Rituximab: Arm 1, Arm 2 = 250 mg/m^2 by vein;
  Arm 1, Arm 2, Arm 3, Arm 4 = 1000 mg/m^2 by vein following Stem Cell Transplant;
  Arm 1, Arm 3 = 375 mg/m² by vein Maintenance Therapy.
  Stem Cell Transplant: Injection of stem cells (Autologous SCT)
- Group 1 - Zevalin + BEAM + Stem Cell Transplant: Zevalin + BEAM + Rituximab Followed by Stem Cell Transplant
  Zevalin: (111In Zevalin) 5 millicurie (mCi) by vein and (90Y Zevalin) 0.4 mCI/kg by vein.
  Carmustine: 300 mg/m^2 by vein.
  Etoposide: 200 mg/m^2 by vein every 12 hours.
  Cytarabine: 200 mg/m^2 by vein every 12 hours.
  Melphalan: 140 mg/m^2 by vein.
  Rituximab: Arm 1, Arm 2 = 250 mg/m^2 by vein;
  Arm 1, Arm 2, Arm 3, Arm 4 = 1000 mg/m^2 by vein following Stem Cell Transplant;
  Arm 1, Arm 3 = 375 mg/m² by vein Maintenance Therapy.
  Stem Cell Transplant: Injection of stem cells (Autologous SCT)
- Group 2 - BEAM + Rituximab + Stem Cell Transplant: BEAM + Rituximab Followed by Stem Cell Transplant and Maintenance Rituximab
  Carmustine: 300 mg/m^2 by vein.
  Etoposide: 200 mg/m^2 by vein every 12 hours.
  Cytarabine: 200 mg/m^2 by vein every 12 hours.
  Melphalan: 140 mg/m^2 by vein.
  Rituximab: Arm 1, Arm 2 = 250 mg/m^2 by vein;
  Arm 1, Arm 2, Arm 3, Arm 4 = 1000 mg/m^2 by vein following Stem Cell Transplant;
  Arm 1, Arm 3 = 375 mg/m² by vein Maintenance Therapy.
  Stem Cell Transplant: Injection of stem cells (Autologous SCT)
- Group 2 - BEAM + Stem Cell Transplant: BEAM + Rituximab Followed by Stem Cell Transplant
  Carmustine: 300 mg/m^2 by vein.
  Etoposide: 200 mg/m^2 by vein every 12 hours.
  Cytarabine: 200 mg/m^2 by vein every 12 hours.
  Melphalan: 140 mg/m^2 by vein.
  Rituximab: Arm 1, Arm 2 = 250 mg/m^2 by vein;
  Arm 1, Arm 2, Arm 3, Arm 4 = 1000 mg/m^2 by vein following Stem Cell Transplant;
  Arm 1, Arm 3 = 375 mg/m² by vein Maintenance Therapy.
  Stem Cell Transplant: Injection of stem cells (Autologous SCT)
Period: Overall Study
Arm/Group | Group 1 - Zevalin + BEAM + Rituximab +Stem Cell Transplant | Group 1 - Zevalin + BEAM + Stem Cell Transplant | Group 2 - BEAM + Rituximab + Stem Cell Transplant | Group 2 - BEAM + Stem Cell Transplant
Started | 6 | 8 | 10 | 6
Completed | 6 | 8 | 9 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Zevalin + BEAM + Rituximab +Stem Cell Transplant | Group 1 - Zevalin + BEAM + Stem Cell Transplant | Group 2 - BEAM + Rituximab + Stem Cell Transplant | Group 2 - BEAM + Stem Cell Transplant | Total
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 7 | 6 | 25
  >=65 years | 1 | 1 | 3 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 4 | 12
  Male | 5 | 5 | 6 | 2 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 0 | 6
  Not Hispanic or Latino | 3 | 5 | 1 | 3 | 12
  Unknown or Not Reported | 0 | 2 | 7 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 10 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 2-Year Progression-Free Survival (PFS)
Description: Response evaluated using the standard criteria response for lymphoma through CT scan.
Time Frame: 2 years (beginning day 30 after treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Zevalin + BEAM + Rituximab +Stem Cell Transplant | Group 1 - Zevalin + BEAM + Stem Cell Transplant | Group 2 - BEAM + Rituximab + Stem Cell Transplant | Group 2 - BEAM + Stem Cell Transplant
Number analyzed (Participants) | 6 | 8 | 10 | 6
Participants | 6 | 8 | 8 | 5

ADVERSE EVENTS:
Time Frame: 3 Years
Arm/Group | Group 1 - Zevalin + BEAM + Rituximab +Stem Cell Transplant | Group 1 - Zevalin + BEAM + Stem Cell Transplant | Group 2 - BEAM + Rituximab + Stem Cell Transplant | Group 2 - BEAM + Stem Cell Transplant
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 1/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 1/10 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 9/10 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Zevalin + BEAM + Rituximab +Stem Cell Transplant (N=6) | Group 1 - Zevalin + BEAM + Stem Cell Transplant (N=8) | Group 2 - BEAM + Rituximab + Stem Cell Transplant (N=10) | Group 2 - BEAM + Stem Cell Transplant (N=6)
CD OTH (Cardiac disorders) | 0 | 0 | 1 | 0
NE OTH (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Group 1 - Zevalin + BEAM + Rituximab +Stem Cell Transplant (N=6) | Group 1 - Zevalin + BEAM + Stem Cell Transplant (N=8) | Group 2 - BEAM + Rituximab + Stem Cell Transplant (N=10) | Group 2 - BEAM + Stem Cell Transplant (N=6)
ALK increased (Investigations) | 1 | 3 | 1/9 | 4
Allergic reaction (Immune system disorders) | 0 | 0 | 1/9 | 1
ALT increased (Investigations) | 0 | 0 | 1/9 | 1
Bacterial (Infections and infestations) | 2 | 2 | 2/9 | 0
Bleeding (no GI no PUL) (Blood and lymphatic system disorders) | 1 | 0 | 0/9 | 0
Bone pain (General disorders) | 0 | 0 | 0/9 | 1
CD OTH (Cardiac disorders) | 0 | 0 | 0/9 | 0
Chest pain (Cardiac disorders) | 0 | 0 | 1/9 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0/9 | 0
Creatinine increased (Investigations) | 0 | 1 | 1/9 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 7 | 4/9 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0/9 | 1
Dysrhythmia (Cardiac disorders) | 0 | 0 | 1/9 | 0
Edema (General disorders) | 0 | 0 | 0/9 | 1
Fatigue (General disorders) | 1 | 0 | 0/9 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 6 | 5/9 | 5
Fever (General disorders) | 0 | 1 | 3/9 | 1
Flu like syndrome (General disorders) | 0 | 0 | 1/9 | 0
Fluid overload (General disorders) | 2 | 2 | 4/9 | 1
Fungal (Infections and infestations) | 0 | 1 | 0/9 | 0
Headache (Nervous system disorders) | 0 | 1 | 1/9 | 0
Hypertension (Vascular disorders) | 2 | 3 | 1/9 | 1
Hypotension (Vascular disorders) | 1 | 1 | 1/9 | 0
IN FEC (Infections and infestations) | 1 | 0 | 0/9 | 0
Nausea (Gastrointestinal disorders) | 6 | 8 | 9/9 | 5
NE COR (Nervous system disorders) | 0 | 0 | 1/9 | 0
NE OTH (Nervous system disorders) | 0 | 0 | 0/9 | 0
Oral mucositis (Gastrointestinal disorders) | 6 | 8 | 7/9 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1/9 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1/9 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2/9 | 2
T bilirubin increased (Investigations) | 1 | 1 | 1/9 | 2
Viral (Infections and infestations) | 1 | 0 | 0/9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT00591630/Prot_SAP_000.pdf